CLINICAL TRIAL: NCT00993148
Title: Maraviroc Plus Darunavir/Ritonavir Study for Treatment-Naïve Patients Infected With R5-tropic HIV-1 Based on Enhanced Sensitivity Trofile
Brief Title: Maraviroc Plus Darunavir/Ritonavir for Treatment-Naïve Patients Infected With R5-tropic HIV-1
Acronym: MIDAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Pfizer (Industry); Tibotec, Inc (Industry)
Responsible Party: Principal Investigator, Babafemi Taiwo, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIDAS
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: HIV-1 Infection; HIV Infections
Keywords: Treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maraviroc plus darunavir/ritonavir (Experimental): Single arm open label trial of maraviroc 150 mg plus darunavir/ritonavir 800/100 mg once daily for 96 weeks
  Interventions: Drug: maraviroc; Drug: darunavir; Drug: ritonavir

INTERVENTIONS:
Drug: maraviroc — 150 mg tab by mouth once daily for 96 weeks
  Other Names: Selzentry
Drug: darunavir — 800 mg tab by mouth once daily for 96 weeks
  Other Names: Prezista
Drug: ritonavir — 100 mg capsule by mouth once daily for 96 weeks
  Other Names: norvir

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a novel combination antiretroviral therapy regimen consisting of maraviroc plus darunavir/ritonavir in treatment-naive patients infected with R5-tropic HIV-1. The hypothesis is that in treatment-naive subjects infected with R5-tropic HIV-1, combination antiretroviral therapy with maraviroc plus darunavir/ritonavir is well tolerated and efficacious.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by any licensed HIV test kit and confirmed by Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA any time prior to study entry
* Plasma HIV-1 RNA 5, 000 to 500,000 copies/mL obtained within 90 days prior to study entry
* Exclusive R5 tropism based on enhanced sensitivity Trofile assay done within 90 days prior to entry
* CD4 cell count > 100 cells/mm3 within 90 days prior to study entry
* HIV genotype (for RT and protease) performed at any time before study entry (Subjects with single or combination NNRTI or NRTI RAM(s) at screening are permitted)
* ARV drug-naïve, defined as no previous ARV treatment at any time prior to study entry
* Negative result from a hepatitis B surface antigen test performed within 90 days prior to study entry
* Negative result from a hepatitis C antibody test performed within 90 days prior to study entry
* Laboratory values obtained within 30 days prior to study entry:

  * ANC >=750/mm3
  * Hemoglobin >=10 g/dL
  * Platelets >=50,000/mm3
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase <=5 x ULN
  * Calculated creatinine clearance (CrCl) >=30 mL/min, as estimated by the Cockcroft-Gault equation*
* Negative serum or urine pregnancy test within 48 hours prior to study entry for women with reproductive potential
* If participating in sexual activity that could lead to pregnancy, the study subjects with reproductive potential must use one form of contraceptive while receiving protocol-specified medications and for 60 days after stopping the medications.
* Men and women age >=18 years
* Ability and willingness of subject or legal guardian/representative to provide informed consent

Exclusion Criteria:

* Serious illness requiring systemic treatment and/or hospitalization until candidate either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to study entry
* Screening HIV genotype obtained any time prior to study entry with any DRV RAM (V11I, V32I, L33F, I47V, I50V, I54L, I54M, T74P, L76V, I84V, and L89V)
* Treatment within 30 days prior to study entry with immune modulators such as systemic steroids, interleukins, interferons, granulocyte colony-stimulating factor (G-CSF), erythropoietin, or any investigational therapy. NOTE: Subjects receiving stable physiologic glucocorticoid doses (defined as prednisone ≤10 mg/day [or equivalent] as a stable or tapering dose) are permitted. Subjects receiving corticosteroids for acute therapy for PCP or asthma exacerbation, or receiving a short course (defined as ≤2 weeks of pharmacologic glucocorticoid therapy) are permitted
* Breast-feeding
* Requirement for any medication that is prohibited with a study medication
* Known allergy/sensitivity to study drugs or their formulations. A history of sulfa allergy is not an exclusion
* Active drug or alcohol use or dependence that could interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babafemi Taiwo, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Quest Clinical Research, San Francisco, California
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - CORECenter, Chicago, Illinois
  - University of Nebraska, Omaha, Nebraska

REFERENCES:
- [Result] Taiwo B, Acosta EP, Ryscavage P, Berzins B, Lu D, Lalezari J, Castro J, Adeyemi O, Kuritzkes DR, Eron JJ, Tsibris A, Swindells S. Virologic response, early HIV-1 decay, and maraviroc pharmacokinetics with the nucleos(t)ide-free regimen of maraviroc plus darunavir/ritonavir in a pilot study. J Acquir Immune Defic Syndr. 2013 Oct 1;64(2):167-73. doi: 10.1097/QAI.0b013e3182a03d95. PMID 23797691

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc + Darunavir/Ritonavir: maraviroc 150 mg plus darunavir/ritonavir 800/100 mg once daily
Period: Overall Study
Arm/Group | Maraviroc + Darunavir/Ritonavir
Started | 25
Completed | 22
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — never initiated treatment | 1

BASELINE CHARACTERISTICS:
Population: HIV-infected treatment naïve participants with R5 virus
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [31 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 15
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 25
Median HIV-1 RNA [Median (Inter-Quartile Range); unit: log 10 copies] — Median HIV-1 RNA
  log 10 copies | 4.62 [4.18 to 4.80]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA >50
Description: Percentage of participants with confirmed plasma HIV-1 RNA > 50 copies/mL
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 24
percentage of participants | 12.5 [2.7 to 32.4]

2. Secondary Outcome: Percentage of Participants With Virologic Failure or Off Study Treatment Regimen
Description: Percentage of participants with virologic failure (confirmed plasma HIV-1 RNA > 50 copies/mL) or off study treatment regimen (composite end point)
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 24
percentage of participants | 12.5 [2.7 to 32.4]

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA >50 Copies/mL
Description: Percentage of participants with confirmed plasma HIV-1 RNA level >50 copies/mL
Time Frame: 48 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 24
percentage of participants | 8.3 [1.0 to 27.0]

4. Secondary Outcome: Signs/Symptoms or Laboratory Toxicities of Grade 3 or Higher
Description: Signs/symptoms or laboratory toxicities of Grade 3 or higher, or of any grade which led to a permanent change or discontinuation of study treatment regimen
Time Frame: 96 weeks
Measure: Number; unit: participants
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 24
participants | 1

5. Secondary Outcome: Drug Resistance Mutations and Co-receptor Tropism Assessed by Trofile ES
Time Frame: At study entry and at the time of virologic failure
Measure: Number; unit: participants
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 24
participants | 0

6. Secondary Outcome: Drug Adherence, Number of Participants With Missed Doses
Description: Drug adherence, assessed as number of participants with missed doses over four-day recall
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 24
participants | 0

7. Secondary Outcome: Trough Concentrations (Ctrough) of Maraviroc
Description: Average trough concentration (Ctrough) of maraviroc
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 24
ng/mL | 39.3 (22.8)

8. Secondary Outcome: Median CD4 Count Change From Baseline
Description: Median changes from baseline in peripheral CD4+ T-cell count
Time Frame: 96 weeks
Measure: Median (Inter-Quartile Range); unit: cells per mm^3
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 24
cells per mm^3 | 247 [119 to 340]

9. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA >50 Copies/mL
Description: Proportion of participants with confirmed plasma HIV-1 RNA level >50 copies/mL
Time Frame: 96 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maraviroc + Darunavir/Ritonavir
Number analyzed (Participants) | 20
percentage of participants | 10 [1.2 to 31.7]

ADVERSE EVENTS:
Arm/Group | Maraviroc + Darunavir/Ritonavir
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No